CLINICAL TRIAL: NCT04952883
Title: A Cross-sectional Study of Endogenous Hydrogen Sulfide and Pulmonary Vascular Remodeling on HRCT in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Hydrogen Sulfide and Pulmonary Vascular Remodeling on HRCT in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2016099
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: The COPD questionnaire was conducted to collect the data of lung function, echocardiography and blood gas analysis, and the pulmonary vessels of HRCT were determined. Blood samples were collected for H2S-related indicators detection.

SUMMARY:
HRCT was used to evaluate pulmonary vascular remodeling in COPD. The role of H2S in pulmonary vascular remodeling in COPD was analyzed, in order to provide a basis for seeking new therapeutic targets.

DETAILED DESCRIPTION:
This study aimed to investigate the relationship between endogenous H2S and pulmonary vascular remodeling on HRCT in patients with COPD through the determination of H2S and its synthase mRNA levels in blood and pulmonary vessels by HRCT, to evaluate the role of H2S in pulmonary vascular remodeling in COPD and to provide a basis for seeking new therapeutic targets. This study had predictive value for clinical prognosis of patients. It had important clinical guiding significance and social and economic benefit to comprehensively understand the pathogenesis of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients meet the GOLD 2016 guidelines for diagnostic criteria of COPD: dyspnea, chronic cough and/or sputum symptoms, exposure to risk factors, and pulmonary function after inhalation of bronchodilator with forced expiratory volume (FEV1)/forced vital capacity (FVC) < 70%.

Exclusion Criteria:

- 1. Other lung diseases such as pneumonia, lung cancer, tuberculosis, pulmonary embolism, heart diseases such as heart failure, ventricular septal defect, patent ductus arteriosus, thoracic deformity and pleural diseases.

2. Patients who are unable to understand and/or complete questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient with stable chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Plasma levels of H2S and its synthase nucleic acid and pulmonary vascular remodeling indexes on HRCT in COPD patients | 1 year

SECONDARY OUTCOMES:
Relationship between plasma H2S and its synthase nucleic acid levels and pulmonary vascular remodeling indexes on HRCT in patients with COPD | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, PHD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided